CLINICAL TRIAL: NCT02966704
Title: A Dual Stable Isotope Method to Assess Dietary Protein Quality in Humans: Characterization of Intrinsically Labelled 15N Milk Protein as a Reference Protein
Brief Title: Stable Isotope Method to Assess Dietary Protein Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL56440.081.16
Record Dates: First submitted 2016-01-08; First posted 2016-11-17 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Biological Availability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- meal 1 (Experimental): mixed meal with high level of intrinsically labeled milk protein
  Interventions: Dietary Supplement: intrinsically labeled milk protein
- meal 2 (Experimental): mixed meal with low level of intrinsically labeled milk protein
  Interventions: Dietary Supplement: intrinsically labeled milk protein

INTERVENTIONS:
Dietary Supplement: intrinsically labeled milk protein

SUMMARY:
The evaluation of protein quality has been identified as the top priority question by the Food and Agricultural Organization (FAO) of the United Nations. However, the current available methods do not precisely estimate protein quality, or need invasive procedures. The proposed 'dual tracer approach' is a non-invasive method to evaluate protein quality in humans.

The present project characterizes the use of 15N-intrinsically-labelled milk protein as a reference-protein for development a non-invasive method that can be used to assess protein quality in human subjects

DETAILED DESCRIPTION:
Rationale: The evaluation of protein quality has been identified as the top priority question by the Food and Agricultural Organization (FAO) of the United Nations. However, the current available methods do not precisely estimate protein quality, or need invasive procedures. The proposed 'dual tracer approach' is a minimal invasive method to evaluate protein quality in humans.

Objective: The present project characterizes the use of 15N-intrinsically-labelled milk protein as a reference-protein for development a minimal invasive method that can be used to assess protein quality in human subjects. For this purpose, our primary objectives are to define the digestive and metabolic behaviour and distribution of the 15N-intrinsically-labelled milk protein compared to the internal standard 13C-spirulina.

Study design: Randomized cross-over trial with two experimental meals. Study population: Healthy male and female, age 18-35y Intervention (if applicable): On two separate test days, subjects will receive a semi liquid meal (pudding) divided in 9 portions, (meal 1: 27 En% Protein,10 En% fat, 62 En% carbohydrates; meal 2: 14 En% Protein,10 En% fat, 75 En% carbohydrates), with intrinsically labelled 15N protein powder. Furthermore, the meal will contain a trace amount of 13C-labelled algae protein as an internal standard. Meals will differ in the amount (e.g. 50g or 25g) of 15N-labelled milk protein.

Main study parameters/endpoints: The ratio of isotopic enrichment (15N/13C) of (total) amino acids of the test meal and the blood plasma as determined by (gas chromatography-) isotope ratio mass spectrometry ((GC)-IRMS).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: A meal challenge with intrinsically labelled protein and addition of stable isotope tracer is frequently used in postprandial studies. Stable isotopes are naturally occurring isotopes and are not harmful for subjects, as there is no decay. Furthermore, placing venous catheters and blood sampling can occasionally cause a local haematoma or bruise and some participants may report pain or discomfort. Subjects have to come to the research facility three times, a screening visit of 1 hour, and 2 experimental days of 7 hours. Subjects will be financially compensated for participation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age: 20 - 35 y
* BMI: 18.5 - 25 kg/m2
* Stable dietary habits
* Veins suitable for cannulation (blood sampling)

Exclusion Criteria:

* Having a history of medical or surgical events that may significantly affect the study outcome
* Medical drug use accept incidental use of paracetamol
* (Chronic) disease which might influence the study outcomes e.g. diabetes mellitus or any other endocrine disorder, active cardiovascular disease, hepatic disease, renal disease, cancer
* Milk protein intolerance
* Alcohol consumption of >14 (women) or > 21 (men) units per week
* Drug abuse
* Moderate intense physical activity (exercise) for more than 5 hours/week
* Reported weight loss or weight gain of > 3 kg in the month prior to pre-study screening
* Reported slimming diet, or medically prescribed diet
* Having a habitual diet with a protein content of <10 En% > 30 En%
* Reported vegan or macrobiotic life-style
* Recent blood donation (<1 month prior to Day 01 of the study)
* Not willing to comply to the controlled dietary intervention guidelines
* Not willing or afraid to give up blood donation during the study
* Personnel of Wageningen University, department of Human Nutrition, their partner and their first and second degree relatives
* Current and within 1 month participation in other research from the Division of Human Nutrition
* Not having a general practitioner

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
ratio of isotopic enrichment | 6 hours

REFERENCES:
- [Derived] van der Wielen N, Khodorova NV, Gerrits WJJ, Gaudichon C, Calvez J, Tome D, Mensink M. Blood 15N:13C Enrichment Ratios Are Proportional to the Ingested Quantity of Protein with the Dual-Tracer Approach for Determining Amino Acid Bioavailability in Humans. J Nutr. 2020 Sep 1;150(9):2346-2352. doi: 10.1093/jn/nxaa205. PMID 32710787